CLINICAL TRIAL: NCT00095459
Title: A Phase I Trial of BAY 43-9006 (Sorafenib) and Bevacizumab in Refractory Solid Tumors With Biologic and Proteomic Analysis
Brief Title: BAY 43-9006 (Sorafenib) and Bevacizumab (Avastin) To Treat Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050022; 05-C-0022; NCT00098592 (obsolete NCT alias)
Record Dates: First submitted 2004-11-04; First posted 2004-11-05 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-04-23

CONDITIONS: Neoplasms
Keywords: Raf-Kinase Inhibitor; Combinatorial Therapy; Pathway Profiling; VEGFR; Bevacizumab; Sorafenib; Advanced Solid Tumors; Angiogenesis; Targeted Therapy; VEGF; Cancer; Solid Tumor; Metastatic Uresectable Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — Bevacizumab; Sorafenib

INTERVENTIONS:
Drug: Bevacizumab
Drug: BAY 43-9006

SUMMARY:
Background:

* BAY 43-9006 is an inhibitor of wild-type and mutant B-Raf and c-Raf kinase isoforms in vitro, but it also inhibits p38, c-kit, VEGFR-2 and PDGFR-Beta affecting tumor growth as well as possibly promoting apoptosis by events downstream of c-Raf.
* Bevacizumab is a humanized IgG1 monoclonal antibody (MAb) that binds all biologically active isoforms of human vascular endothelial growth factor (VEGF, or VEGF-A) with high affinity (k(d)= 1.1nM)
* The most common adverse events associated with bevacizumab of any severity include asthenia, pain, headache, hypertension, diarrhea, stomatitis, constipation, epistaxis, dyspnea, dermatitis and proteinuria.
* This Phase I trial is open to patients with all solid tumors.

Objectives:

* Determine the safety and toxicity of the combination of BAY 43-9006 (Sorafenib) and bevacizumab.
* Determine estimates of biochemical changes in the Ras-Raf-MAPK and VEGF signal transduction pathways in tumor and stromal cells in response to treatment at the MTD, at least in a pilot fashion, if those changes are statistically significant.

Eligibility:

* Adults with histologically documented solid tumor malignancy that is metastatic or unresectable and for which standard curative therapies do not exist or are no longer effective.
* Patients must be off prior chemotherapy, radiation therapy, hormonal therapy, or biological therapy for at least 4 weeks.
* All patients enrolling in cohort 2 must have at least one lesion amenable to biopsy.
* ECOG performance status 0 or 1 and adequate organ and marrow function.

Design:

* Cohort I will receive BAY 43-9006 and bevacizumab together at the start of study in a dose escalation fashion.
* Cohort II will be randomized as to which agent they receive for cycle one. Cycles 2 and beyond are treated using both agents.
* Tumor biopsies will be obtained from patients in Cohort II before treatment, two weeks into mono-therapy, and two weeks into combinatorial therapy.
* DCE-MRI studies will be obtained on patients in Cohort II before treatment, two weeks into monotherapy, four weeks into monotherapy, and two weeks into combinatorial therapy.
* FDG-PET studies will be obtained on patients in Cohort II before treatment, two weeks into mono-therapy, and two weeks into combinatorial therapy.
* Patients will be evaluated for toxicity in clinic every 2 weeks for Cycles 1 and 2, and then every 4 weeks.
* Patients will be evaluated for response every 8 weeks using the RECIST criteria.
* Approximately 62 patients will be needed to achieve the objectives of the trial.

DETAILED DESCRIPTION:
Background:

* BAY 43-9006 is an inhibitor of wild-type and mutant B-Raf and c-Raf kinase isoforms in vitro, but it also inhibits p38, c-kit, VEGFR-2 and PDGFR-Beta affecting tumor growth as well as possibly promoting apoptosis by events downstream of c-Raf.
* Bevacizumab is a humanized IgG1 monoclonal antibody (MAb) that binds all biologically active isoforms of human vascular endothelial growth factor (VEGF, or VEGF-A) with high affinity (k(d)= 1.1nM)
* The most common adverse events associated with bevacizumab of any severity include asthenia, pain, headache, hypertension, diarrhea, stomatitis, constipation, epistaxis, dyspnea, dermatitis and proteinuria.
* This Phase I trial is open to patients with all solid tumors.

Objectives:

* Determine the safety and toxicity of the combination of BAY 43-9006 (Sorafenib) and bevacizumab.
* Determine estimates of biochemical changes in the Ras-Raf-MAPK and VEGF signal transduction pathways in tumor and stromal cells in response to treatment at the MTD, at least in a pilot fashion, if those changes are statistically significant.

Eligibility:

* Adults with histologically documented solid tumor malignancy that is metastatic or unresectable and for which standard curative therapies do not exist or are no longer effective.
* Patients must be off prior chemotherapy, radiation therapy, hormonal therapy, or biological therapy for at least 4 weeks.
* All patients enrolling in cohort 2 must have at least one lesion amenable to biopsy.
* ECOG performance status 0 or 1 and adequate organ and marrow function.

Design:

* Cohort I will receive BAY 43-9006 and bevacizumab together at the start of study in a dose escalation fashion.
* Cohort II will be randomized as to which agent they receive for cycle one. Cycles 2 and beyond are treated using both agents.
* Tumor biopsies will be obtained from patients in Cohort II before treatment, two weeks into mono-therapy, and two weeks into combinatorial therapy.
* DCE-MRI studies will be obtained on patients in Cohort II before treatment, two weeks into monotherapy, four weeks into monotherapy, and two weeks into combinatorial therapy.
* FDG-PET studies will be obtained on patients in Cohort II before treatment, two weeks into mono-therapy, and two weeks into combinatorial therapy.
* Patients will be evaluated for toxicity in clinic every 2 weeks for Cycles 1 and 2, and then every 4 weeks.
* Patients will be evaluated for response every 8 weeks using the RECIST criteria.
* Approximately 62 patients will be needed to achieve the objectives of the trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have a solid tumor malignancy that is metastatic or unresectable and for which standard curative therapies do not exist or are no longer effective.

Patients must have histological documentation of cancer confirmed in the Laboratory of Pathology/NCI.

Patients must be off prior chemotherapy, radiation therapy, hormonal therapy, or biological therapy for at least 4 weeks. Patients who were receiving mitomycin C, nitrosoureas, or carboplatin must be 6 weeks from the last administration of chemotherapy. Patients with prostate cancer must continue to receive LHRH agonist (unless orchiectomy has been performed). Patients should not be receiving complementary/alternative therapy while on study. Furthermore, complementary therapy should be stopped at least 7 days prior to enrollment. Any patient who has undergone therapy with a monoclonal antibody must be at least 8 weeks from the last treatment.

All patients enrolling in cohort 2 must have at least one lesion amenable to biopsy. This determination will be made by a member of the interventional radiology team or surgical associate investigator and an associate investigator. This requirement is not necessary for patients in cohort 1.

Age greater than 18 years.

ECOG performance status 0 or 1.

Life expectancy of greater than 3 months.

Patients must have adequate organ and marrow function as defined below:

* Leukocytes greater than 3,000/microliter
* Absolute neutrophil count greater than 1,200/microliter

Platelets greater than 100,000/microliter

* Total Bilirubin less than or equal to 1.5 times the institutional upper limits of normal
* AST(SGOT) and ALT(SGPT) less than or equal to 2.5 times the institutional upper limit of normal
* Creatinine less than or equal to 1.5 mg/dL OR creatinine clearance greater than 45 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.
* Activated partial thromboplastin time (PTT) less than 1.25 times the institutional upper limits of normal
* Prothrombin Time (PT) OR INR less than 1.25 times the institutional upper limits of normal
* Amylase and Lipase less than or equal to the institutional upper limit of normal
* Spot Urine Protein Creatinine Ratio less than 0.5; If result is 0.5 or more, a 24-hour urine for protein excretion must be less than 1000mg

Patients must have recovered from toxicity related to prior therapy to at least CTEP grade 1 (defined by CTC 3.0). Chronic stable grade 2 peripheral neuropathy secondary to neurotoxicity from prior therapies may be considered on a case by case basis by the Principal Investigator.

Women of child-bearing potential and men must agree to use adequate contraception (abstinence; hormonal or barrier method of birth control) for the study and at least 2 months after completion. Pregnant women will not be eligible for study.

Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Brain metastases

* Patients who have a history of remote CNS metastases that have undergone "curative therapy" by radiation therapy, gamma knife therapy, or surgery and have remained without recurrence for a period of greater than or equal to 2 years will be considered on a case-by-case basis.
* CNS imaging will not be mandated for all patients. However, if there is clinical suspicion of CNS involvement, a contrast CT or MRI of the brain will be required. Screening CNS scans should be required for certain tumor types with relatively high risk of CNS metastases, including but not limited to melanoma, RCC, breast, lung.

Thrombotic or embolic events within the past 6 months such as a cerebrovascular accident (including transient ischemic attacks), pulmonary embolism, unstable angina, or myocardial infarction.

Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (AHA Class II or worse), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

-Patients with evidence of active infection will become eligible for reconsideration 7 days after completing antibiotic therapy.

HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with BAY 43-9006, bevacizumab, and/or the combination.

Patients who have been treated with BAY 43-9006 or bevacizumab will be excluded

Hypertension defined as systolic blood pressure greater than 140 mmHg or diastolic pressure greater than 90 mmHg despite optimal medical management.

Proteinuria defined as a 24-hour urine protein excretion greater than 1000 mg. Spot urine analysis for protein creatinine ratio (UPC) of 0.5 or greater will require a 24-hour urine to determine eligibility for enrollment.

Therapeutic anticoagulation with coumadin, heparins, or heparinoids.

Serious non-healing wounds (including wounds healing by secondary intention), acute or non-healing ulcers, or bone fractures within 3 months of fracture. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abcesses within 28 days will be excluded.

Evidence of bleeding diathesis

Impairment of swallowing that would preclude administration of BAY 43-9006.

History of hemoptysis or surgery within the past 28 days.

Patients with squamous cell carcinoma of the lungs will be excluded due to risk of fatal pulmonary hemorrhage. If a patient has a history of any type primary lung cancer and hemoptysis, they will be excluded.

History of high grade varices.

Use of herbal supplements are not permitted within 14 days of trial commencement and on study. Vitamin supplement (above a typical single multi-vitamin) usage is discouraged unless clearly indicated by an existing medical condition. An Associate or Principal Investigator will have the discretion regarding which vitamin supplements are permitted.

Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2004-11-02; Primary Completion 2005-11-01 (Actual); Study Completion 2012-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elise C Kohn, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Campbell SL, Khosravi-Far R, Rossman KL, Clark GJ, Der CJ. Increasing complexity of Ras signaling. Oncogene. 1998 Sep 17;17(11 Reviews):1395-413. doi: 10.1038/sj.onc.1202174. PMID 9779987
- [Background] Cohen Y, Xing M, Mambo E, Guo Z, Wu G, Trink B, Beller U, Westra WH, Ladenson PW, Sidransky D. BRAF mutation in papillary thyroid carcinoma. J Natl Cancer Inst. 2003 Apr 16;95(8):625-7. doi: 10.1093/jnci/95.8.625. PMID 12697856
- [Background] Chong H, Vikis HG, Guan KL. Mechanisms of regulating the Raf kinase family. Cell Signal. 2003 May;15(5):463-9. doi: 10.1016/s0898-6568(02)00139-0. PMID 12639709